CLINICAL TRIAL: NCT06145893
Title: A Phase III Clinical Study of Efficacy and Safety of Hemay005 Tablets in Patients With Behçet's Disease
Brief Title: A Study of Efficacy and Safety of Hemay005 Tablets in Patients With Behçet's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HM005BD3S01
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: Behçet's Disease
Keywords: Behçet's Disease
MeSH Terms: conditions — Behcet Syndrome | interventions — Hemay005; Cyclic Nucleotide Phosphodiesterases, Type 4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hemay005 high dose group (Experimental): In Core-treatment period, subject will take Hemay005 60mg twice daily for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 60mg twice daily for 40 weeks.
  Interventions: Drug: Hemay005
- Hemay005 lower dose group (Experimental): In Core-treatment period, subject will take Hemay005 45mg twice daily for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 45mg twice daily for 40 weeks.
  Interventions: Drug: Hemay005
- Placebo (Placebo Comparator): In Core-treatment period, subject will take placebo for 12 weeks, and in the following extend-treatment period, subject will take Hemay005 60mg or hemay005 45mg twice daily according to pre-allocation at randomization visit for 40 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemay005 — Hemay005 tables 60mg bid p.o;
  Other Names: Mufemilast; Phosphodiesterase 4 (PDE4) inhibitors
  Arms: Hemay005 high dose group
Drug: Hemay005 — Hemay005 tables 45mg bid p.o;
  Other Names: Mufemilast; Phosphodiesterase 4 (PDE4) inhibitors
  Arms: Hemay005 lower dose group
Drug: Placebo — placebo to Hemay005 tables bid p.o
  Arms: Placebo

SUMMARY:
This is a phase 3, multi-center, randomized, placebo-controlled, double-blind, parallel-group study with an equal randomization among the Hemay005 high dose, lower dose and placebo treatment groups. After subject randomization, each subject will enter an core-treatment Phase for 12 weeks following an extended-treatment phase for another 40 weeks and a follow up phase for 4weeks.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-parallel controlled phase III clinical study. The study consists of four phases, namely the screening period, the core treatment period, the extension period, and the drug discontinuation observation period.

Screening period: All subjects will undergo a screening period for up to 8 weeks prior to the baseline visit (V2, randomization day, Day 0).

Core treatment period: Patients with Behçet's disease (BD) meeting the eligibility criteria upon screening will be randomized in a 1:1: 1 ratio to the Hemay005 Tablets 45 mg BID test group, Hemay005 Tablets 60 mg BID test group, or the placebo group. They will first be given escalating doses for 7 days; subsequently starting from Day 7, they will be given Hemay005 Tablets 45 mg BID or 60 mg BID or the placebo BID continuously until Week 12.

Extension period: Considering benefits for subjects in the placebo group, and to observe the efficacy and safety of long-term treatment, all subjects will enter a 40-week extension period at the end of the core treatment period. Subjects enrolled in the test groups for the core treatment period will continue treatment at the dose for the core treatment period for 40 weeks during the extension period. Subjects enrolled in the placebo group for the core treatment period will be randomized in a 1:1 ratio during the extension period to either the Hemay005 Tablets 45 mg BID test group or Hemay005 Tablets 60 mg BID test group for treatment for 40 weeks. For the first week of extended treatment, subjects previously enrolled in the placebo group will need to undergo the same dose titration phase as for the core treatment period (Days 0-6), so that the same dosing schedule as for the two treatment groups would be achieved by the 7th day, in an effort to mitigate the intolerabilities such as gastrointestinal reactions, thus further protecting subjects' safety. If, during the dose titration phase of the extension period or during extended treatment, the subject cannot tolerate the prescribed dose, this will be handled at the investigator's discretion using the same method as for the core treatment period.

Drug discontinuation observation period: All subjects in the study (including those who prematurely discontinued treatment for any reason) will be observed for 4 weeks following the end of the last study dose.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and voluntarily signing the Informed Consent Form (ICF) for this study;
2. Age 18-75 years (inclusive), male or female;
3. Diagnosed as BD based on the ICBD-2013;
4. At least 2 oral ulcers present at V1 (screening), and:

   1. at least 2 oral ulcers present at V2 (the day of randomization) when V2 occurs 14-56 days after V1; OR
   2. at least 3 oral ulcers present at V2 (the day of randomization) when V2 occurs 0-13 days after V1;
5. Applicability of systemic treatment for oral ulcers: Based on the severity of the disease and the involved area, the investigator determines that the patient's oral ulceration is not suitable for topical treatment or that the patient's oral ulceration cannot be effectively controlled by topical treatment, so that systemic treatment is to be used;
6. Throughout the study period from signing of ICF through 3 months after the last study dose, women of childbearing potential and male subjects who have not undergone vasoligation should use effective contraceptive measures, including vasoligation, abstinence, intrauterine device (IUD), hormones (oral, patches, rings, injections, implants) and barrier methods (diaphragms, cervical caps, sponges, condoms);
7. Being able to comply with the follow-up schedule and other protocol requirements.

Exclusion Criteria:

1. Active lesions associated with BD in major organs requiring immunosuppressive treatment, e.g., those in lungs (e.g., pulmonary aneurysm), blood vessels (e.g., thrombophlebitis, recurrent malignant aneurysms), gastrointestinal tract (e.g., gastrointestinal ulcers), and central nervous system (e.g., meningoencephalitis); Note: Patients with refractory BD who experienced gastrointestinal perforation, active bleeding, or obstruction, etc. within 3 months prior to randomization are to be excluded.
2. Any clinically significant heart disease (including but not limited to: unstable ischemic heart disease, NYHA III/IV left ventricular failure, or myocardial infarction) or clinically significant 12-lead ECG abnormalities detected during the 6 months prior to screening, which, at the investigator's discretion, may put the subject at safety risk or may interfere with the study assessments;
3. Use of the following immunomodulatory therapies:

   * Colchicine within 7 days prior to randomization;
   * Perazathioprine, mycophenolate, baritinib, or tofacitinib within 10 days prior to randomization;
   * Cyclosporine, methotrexate, cyclophosphamide, thalidomide, or dapsone within 4 weeks (28 days) prior to randomization;
   * Biologics within 5 half-lives prior to randomization, e.g.:

     * Etanercept within 4 weeks prior to randomization;
     * Infliximab or leflunomide within 8 weeks prior to randomization;
     * Adalimumab, golimumab, abatacept, or tolizumab within 10 weeks prior to randomization;
     * Secukinumab within 6 months prior to randomization;
4. Intraarticular or systemic corticosteroid treatment prior to randomization and within 5 pharmacokinetic/pharmacodynamic half-lives; Note: For subjects with eye symptoms, glucocorticoid eye drops are allowed throughout the trial (except for within 24 hours prior to a trial visit).
5. Chinese patent medicines with immunomodulatory effect within 2 weeks prior to randomization; any Chinese pate nt medicines or decoctions within 2 weeks prior to randomization that might affect efficacy evaluation, or containing sinomenine, total glucoside of paeony, or tripterygium wilfordii, etc.;
6. Laboratory tests:

   * Hemoglobin ≤85g/L;
   * White blood cell count <3.0×10^9/L or >14×10^9/L;
   * Platelets <100×10^9/L;
   * Serum creatinine >1.5 mg/dL (>132.6 μmol/L);
   * Total bilirubin of >2.0 mg/dL (>34.2 μmol/L);
   * Both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥1.5×ULN; Note: The above tests can be repeated at most once during the screening period. If the result within 2 weeks prior to randomization falls into the specified range, the subject is eligible for the study;
7. Use of potent inducers of cytochrome P450 enzymes (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin sodium) within 4 weeks prior to randomization;
8. Other autoimmune diseases or chronic inflammatory diseases associated with immunity, e.g., rheumatic fever, rheumatoid arthritis, systemic lupus erythematosus, dermatomyositis, multiple sclerosis, Sjögren's syndrome, and inflammatory bowel disease;
9. Currently active infections or recurrent bacterial, fungal, viral, mycobacterial or other infectious diseases (including but not limited to tuberculosis, atypical mycobacteriosis, hepatitis B, hepatitis C, herpes zoster, histoplasmosis, and coccidiosis; however, onychomycosis is excluded), which, at the investigator's discretion, may put the subject at safety risk; Note: Subjects positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody, or with a history of active mycobacterial infection of any species (including Mycobacterium tuberculosis) within 3 years prior to screening visit should be excluded. Screening is permitted if the subject has been cured for at least 3 years prior to randomization with documentation available for verification;
10. Clinically significant chest X-ray or CT abnormalities, which, at the investigator's discretion, may put the subject at safety risk; Note: If a chest X-ray or CT was performed within 3 months prior to V1, the examination may be omitted for V1;
11. History of transplantation or immunodeficiency;
12. Positive for human immunodeficiency virus (HIV) antibody or treponema pallidum antibody test;
13. Currently having a malignant tumor, or a history of any malignant tumor within 5 years prior to screening (except for treatment-experienced squamous cell carcinoma in situ of the skin, basal cell carcinoma or cervical carcinoma in situ with no evidence of relapse within the past 12 months);
14. Use of any clinical investigational product within 4 weeks prior to randomization or 5 pharmacokinetic/pharmacodynamic half-lives, whichever is longer; Note: Subjects who have participated in HM005BD2S01 study are not eligible to participate in this trial;
15. Known allergy to the study drug or any of its components or allergic constitution;
16. A history of alcohol or drug abuse or dependence, or psychiatric disorder;
17. Any conditions that may interfere with oral drug absorption, e.g., subtotal gastrectomy, clinically significant diabetic gastrointestinal disease, or certain types of bariatric surgery such as gastric bypass surgery, not including procedures that simply separate the stomach into separate chambers such as gastric banding surgery;
18. Prior use of apremilast;
19. Female subjects who are pregnant or breast feeding;
20. Concomitant serious, progressive, or uncontrolled diseases, with which participation in the study may, at the investigator's discretion, put the subject at potential risk or affect the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessed by oral ulcers | week 12
  Area under the curve (AUC) of the number of oral ulcers in BD patients from baseline to Week 12

SECONDARY OUTCOMES:
efficacy assessed by oral ulcers | week 12, 22, 32, 42, 52
  Complete response rate for oral ulcers at Week 12，22，32，42，52; A complete response is defined as the proportion of subjects who are oral ulcer free
pain of oral ulcers assessed by VAS | week 12, 22, 32, 42, 52
  Change from baseline in the pain of oral ulcers as measured by VAS at Week 12，22，32，42，52
efficacy assessed by genital ulcers | week 12, 22, 32, 42, 52
  Complete response rate for genital ulcers at Week 12，22，32，42，52 for subjects who had genital ulcers at Baseline; A complete response is defined as the proportion of subjects who are genital ulcer-free
pain of genital ulcers assessed by VAS | week 12, 22, 32, 42, 52
  Change from baseline in the pain of genital ulcers, as measured by VAS at Week 12，22，32，42，52 in subjects who had genital ulcers at baseline
efficacy assessed by BDCAF | week 12, 22, 32, 42, 52
  Change from baseline in disease activity as measured by Behçet's Disease Current Activity scores (BD Current Activity Form) at Week 12，22，32，42，52
efficacy assessed by BSAS | week 12, 22, 32, 42, 52
  Change from Baseline in Behçet's Syndrome Activity Score (BSAS) at Week 12，22，32，42，52
efficacy assessed by oral ulcers | week 1, 2, 4, 6, 8, 10, 12
  Time to oral ulcer resolution (complete response), ie, the first instance when a subject has a complete response, during the Placebo-controlled Treatment Phase
efficacy assessed by oral ulcers | week 1, 2, 4, 6, 8, 10, 12
  Proportion of subjects with no oral ulcers following complete response, ie, the first time when a subject has a complete response, during the Placebo-controlled Treatment Phase
efficacy assessed by oral ulcers | week 1, 2, 4, 6, 8, 10, 12
  Number of oral ulcers following loss of complete response, ie, the first instance when a subject has a reappearance of oral ulcers following a complete response, during the Placebo-controlled Treatment Phase
efficacy assessed by oral ulcers | week 1, 2, 4, 6, 8, 10, 12
  Time to recurrence of oral ulcers following loss of complete response, ie, the first instance when a subject has a reappearance of oral ulcers following a complete response, during the Placebo-controlled Treatment Phase
efficacy of skin lesions assessed by PGA score | week 12, 22, 32, 42, 52
  Change from baseline in the total score of the Static Physician's Global Assessment (PGA) of skin lesions (acne-like lesions, folliculitis and erythema nodosum) of BD at Week 12，22，32，42，52 in subjects who had BD skin lesions at baseline
efficacy assessed by oral ulcers | week 2, 4, 6, 8, 10, 12
  Proportion of subjects achieving an oral ulcer complete response (oral ulcer-free) by Week 6, after start of dosing, and who remain oral ulcer free for at least 6 additional weeks during the 12-week Placebo-controlled Treatment Phase
Quality of life measured by BD QoL | week 12, 22, 32, 42, 52
  Change from baseline in the BD QoL score at Week 12，22，32，42，52
Quality of life measured by SF-36 | week 12, 22, 32, 42, 52
  Change from baseline in SF-36 score at Week 12, 22，32，42，52
efficacy assessed by tender and/or swollen joints | week 12, 22, 32, 42, 52
  Change from baseline in number of tender and/or swollen joints associated with BD at Week 12，22, 32, 42, and 52 in subjects who had BD-related tender and/or swollen joints at baseline;
efficacy assessed by gastrointestinal activity | week 12, 22, 32, 42, 52
  Changes from baseline in Disease Activity Index for Intestinal Behçet's Disease (DAIBD) score at Weeks 12, 22, 32, 42, and 52
efficacy assessed by gastrointestinal symptoms | week 1, 12, 52
  Changes from baseline in Global GI symptoms assessment at Weeks 12 and 52
efficacy assessed by biomarkers. | week 12, 22, 32, 42, 52
  Changes from baseline in CRP and ESR at Weeks 12, 22, 32, 42, and 52;
efficacy assessed by eye symptoms. | week 12, 22, 32, 42, 52
  Changes from baseline in best corrected visual acuity (BCVA) at Weeks 12, 22, 32, 42, and 52, and changes from baseline in improvement of inflammation (slit lamp and/or ophthalmoscopy/fundus photography optical coherence tomography (OCT), etc.) at Weeks 12 and 52
population pharmacokinetics (PopPK) | week 4, 12
  Area under the curve (AUC)
population pharmacokinetics (PopPK) | week 4, 12
  Maximum Plasma Concentration (Cmax)
population pharmacokinetics (PopPK) | week 4, 12
  Minimum Plasma Concentration (Cmin)
population pharmacokinetics (PopPK) | week 4, 12
  Time to peak (Tmax)
population pharmacokinetics (PopPK) | week 4, 12
  Elimination half-life (T1/2)
population pharmacokinetics (PopPK) | week 4, 12
  Clearance (Cl)
safety assessed by Type, frequency, severity and relationship with drug of AEs | week 1, 2, 4, 6, 8, 10, 12, 22, 32, 43, 52, 56
  Type, frequency, severity and relationship with Hemay005 of AEs
safety and tolerability assessed by discontinuation due to AEs | week 1, 2, 4, 6, 8, 10, 12, 22, 32, 43, 52, 56
  Number of subjects prematurely discontinuing the investigational product due to AE
safety and feasibility assessed by lab examinations | week 1, 2, 4, 6, 8, 10, 12, 22, 32, 43, 52, 56
  Frequency of clinically significant changes in vital signs, weight, laboratory findings, physical examination, and/or 12-lead ECG

OTHER OUTCOMES:
efficacy assessed by oral and genital ulcers | week 12
  The AUC for the combined number of oral and genital ulcers from baseline through Week 12
efficacy assessed by genital ulcers | week 1, 2, 4, 6, 8, 10, 12
  Time to genital ulcer complete response, ie, the first instance when a subject has a complete response, during the Placebo-controlled Treatment Phase
efficacy assessed by genital ulcers | week 1, 2, 4, 6, 8, 10, 12
  Proportion of subjects with no genital ulcers following complete response, ie, the first time when a subject has a complete response, during the Placebo-controlled Treatment Phase
efficacy assessed by genital ulcers | week 1, 2, 4, 6, 8, 10, 12
  Number of genital ulcers following loss of complete response ie, the first instance when a subject has a reappearance of oral ulcers following a complete response, during the Placebo-controlled Treatment Phase

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Doctor, Principal Investigator — Peking University People's Hospital
Locations (22):
- China (22):
  - Beijing Friendship hospital capital medical hospital, Beijing, Beijing Municipality
  - Peking university first hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality
  - Xuanwu hospital capital medical university, Beijing, Beijing Municipality
  - The first affiliated hospital of Xiamen University, Xiamen, Fujian
  - Guangdong second provincial central hospital, Guangzhou, Guangdong
  - Sun Yat-Sen memorial hospital, Guangzhou, Guangdong
  - The third affiliated hospital sun yat-sen university, Guangzhou, Guangdong
  - The university of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated hospital of Guilin Medical university, Guilin, Guangxi
  - The second hospital of Hebei medical university, Shijiazhuang, Hebei
  - Xinxiang Central hospital, Xinxiang, Henan
  - The first affiliated hospital of Nanchang university, Nanchang, Jiangsu
  - The first affiliated hospital of Soochow university, Suzhou, Jiangsu
  - The affiliated hospital of Xuzhou medical university, Xuzhou, Jiangsu
  - Jilin Province People's hospital, Changchun, Jilin
  - Linyi People's Hospital, Linyi, Shandong
  - Tongji hospital of Tongji university, Shanghai, Shanghai Municipality
  - Second hospital of shanxi medical university, Taiyuan, Shanxi
  - The first affiliated hospital, Zhejiang University school of medicine, Hangzhou, Zhejiang
  - The first affiliated hospital of Wenzhou Medical university, Wenzhou

IPD SHARING:
Plan to Share IPD: No